CLINICAL TRIAL: NCT04056715
Title: Extended Ambulatory Monitoring With iRhythm Zio XT Improves Care of Patients With Hypertrophic Cardiomyopathy
Brief Title: Extended ECG Monitoring in HCM Patients
Acronym: EXAMINE-HCM
Status: Completed | Type: Observational
Sponsor: iRhythm Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: iRT-001-2019
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hypertrophic Cardiomyopathy; Nonsustained Ventricular Tachycardia; Ventricular Tachycardia; Atrial Fibrillation; Arrhythmia
Keywords: electrocardiography; electrocardiogram; mobile cardiac monitoring; ambulatory monitoring; ECG; EKG
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Tachycardia, Ventricular; Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HCM Group: Eligible HCM subjects will be monitored for arrhythmias with a 2-week ECG patch.
  Interventions: Device: Zio XT

INTERVENTIONS:
Device: Zio XT — ambulatory cardiac monitoring device

SUMMARY:
The purpose of this study is to determine, among a large cohort of 300 consecutive patients with hypertrophic cardiomyopathy, if extended ambulatory monitoring using the iRhythm Technologies, Inc. Zio XT device results in identifying a greater burden of nonsustained ventricular tachyarrhythmia (nsVT) compared to current ACCF/AHA guideline recommended 48-hour monitoring.

DETAILED DESCRIPTION:
Optimal duration to monitor patients for identifying nsVT remains unclear. The investigators aim to determine the prevalence and burden of nsVT with longer term monitoring with the iRhythm Zio XT device over a 2-week period vs. 48 hours; and whether, this greater burden of nsVT compared to conventional shorter monitoring potentially identifies a subset of HCM patients who may be at higher risk of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age at time of informed consent and must not be a member of a vulnerable population.
* Subject has been diagnosed with hypertrophic cardiomyopathy, as defined by a maximal LV wall thickness of ≥15 mm anywhere in LV wall, in absence of another cause that could be responsible for the LV hypertrophy.
* Subject eligible to receive the Zio XT device per the current approved indications for use.

Exclusion Criteria:

* Subject with pacemaker
* Known skin allergies or reaction to adhesives
* The investigator deems a condition that could limit a subject's ability or unwillingness to participate in the study, comply with study required monitoring and/or follow-up visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the hypertrophic cardiomyopathy population will be recruited.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Total number of nsVT runs through 14 days of ambulatory cardiac monitoring, as compared to the first 48 hours. | 14 days
  Compare the number of nsVT runs detected between the first 48 hours vs 2 weeks of ambulatory cardiac monitoring.

SECONDARY OUTCOMES:
Total number of atrial fibrillation runs through 14 days of ambulatory cardiac monitoring, as compared to the first 48 hours. | 14 days
  Compare the number of AF runs detected between the first 48 hours vs 2 weeks of ambulatory cardiac monitoring.
Number of clinical management decisions based on 14 days of ambulatory cardiac monitoring, as compared to the first 48 hours ambulatory cardiac monitoring. | 14 days
  Compare the number clinical decisions based on the first 48 hours vs 14 days of ambulatory cardiac monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Maron, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No